CLINICAL TRIAL: NCT04329975
Title: Specified Drug Use-results Survey (Long-term Use) on MINIRINMELT® OD Tablet 25μg / 50μg in Treatment for Male Nocturia Due to Nocturnal Polyuria
Brief Title: Specified Drug Use-results Survey (Long-term Use) on MINIRINMELT® OD Tablet (Nocturia)
Acronym: NOC01
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000346
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Nocturia Due to Nocturnal Polyuria
Keywords: Hyponatremia; Long-term treatment
MeSH Terms: conditions — Hyponatremia | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Nocturia: Participants with nocturia due to nocturnal polyuria treated with MINIRINMELT OD Tablet 25μg or 50μg as per daily clinical practice.
  Interventions: Drug: Desmopressin

INTERVENTIONS:
Drug: Desmopressin — Desmopressin (MINIRINMELT OD tablet) 25μg or 50μg, orally.
  Other Names: MINIRINMELT

SUMMARY:
To investigate the incidence and risk factors of desmopressin-induced hyponatremia during long-term treatment (1 year [52 weeks]) of MINIRINMELT orally disintegrating (OD) tablets 25μg/50μg (drug) for nocturia caused by nocturnal polyuria in men in daily clinical practice, and to confirm the compliance with proper use of this drug in clinical practice and to investigate the effectiveness of risk minimization activities.

ELIGIBILITY:
Inclusion Criteria:

* Participants who received the MINIRINMELT for the first time in men with nocturia due to nocturnal polyuria, an indication for drug.

Exclusion Criteria:

* No exclusion criteria defined for this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who received the MINIRINMELT for the first time in men with nocturia due to nocturnal polyuria, an indication for drug.
Sampling Method: Non-Probability Sample
Enrollment: 1087 (Actual)
Dates: Start 2020-05-19 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Occurrence of Hyponatremia | 1 year
  Hyponatremia will be confirmed by the investigator if the serum sodium value is 130 mmol/L or less.
Time to Onset of Hyponatremia | 1 year
Distribution of Serum Sodium Levels | 1 year
  Number of participants with mild decrease (serum sodium 134-130 mmol/L); moderate decrease (serum sodium <130 mmol/L) and severe decrease (serum sodium <=125 mmol/L) in serum sodium levels will be presented.
Factors Affecting the Occurrence of Desmopressin-induced Hyponatremia | 1 year
  To evaluate the role of the following factors in the study: adverse drug reactions (ADRs) incidence rate by background factors such as dose of MINIRINMELT 25 or 50 μg, participant age, baseline serum sodium levels, kidney function according to creatinine clearance, medical history and concomitant medications.

SECONDARY OUTCOMES:
Onset Situation of Adverse Drug Reaction/Infectious Disease | 1 year
  An adverse event (AE) is any untoward medical occurrence that did not necessarily have a causal relationship with MINIRINMELT 25 or 50 μg.
  An ADR is an AE evaluated by the Investigator as being probably or possibly causally related to treatment with the MINIRINMELT 25 or 50 μg.
Onset Situation of Serious Adverse Events (SAEs) | Up to 1 year
  A SAE is any event that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity or congenital anomaly/birth defect or was an important medical event that could have jeopardized the participant's safety or required medical or surgical intervention to prevent 1 of the outcomes listed above.
Factors Affecting Safety | 1 year
  To evaluate the role of the following factors in the study: adverse drug reactions incidence rate by background factors such as dose of MINIRINMELT 25 or 50 μg, participant age, baseline serum sodium levels, kidney function according to creatinine clearance, medical history and concomitant medications.
Compliance with proper use of drug | 1 year
  Number of participants with proper use of drug (MINIRINMELT 25 or 50 μg) will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (1):
- Survey Site (there may be other sites in this country), Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No